CLINICAL TRIAL: NCT06679283
Title: Surgical Treatment of Peri-implantitis With Adjunctive Application of Platelet Rich Fibrin (PRF) Compared With Open Flap Debridement (OFD) Alone: A 12-month Randomised Clinical Trial
Brief Title: Surgical Treatment of Peri-implantitis With Adjunctive Application of Platelet Rich Fibrin (PRF)
Acronym: PRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRF
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Peri-Implantitis; Bone Resorption; Platelet-Rich Fibrin
Keywords: platelet rich fibrin, peri-implantitis
MeSH Terms: conditions — Peri-Implantitis; Bone Resorption | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Intervention Model Description: Parallel armed, randomised, single-blinded, controlled, clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcome measures are being assessed by a clinician blinded to the patient allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open flap debridement with a chemo-electric device + PRF (Experimental): A mucoperiosteal flap will be raised to visualize the peri-implant defect, granulation tissue will be removed and the implant surface will be cleaned with a chemo-electric device. Thereafter venous blood will be taken, PRF clots and membranes will be prepared after blood centrifugation. The clots and membrane will be applied into the defect. Finally the flap is closed.
  Interventions: Procedure: Open flap debridement with a chemo-electric device + PRF
- Open flap debridement with a chemo-electric device alone (Active Comparator): A mucoperiosteal flap will be raised to visualize the peri-implant defect, granulation tissue will be removed and the implant surface will be cleaned with a chemo-electric device. Thereafter the flap is closed.
  Interventions: Procedure: Open flap debridement with a chemo-electric device alone (control)

INTERVENTIONS:
Procedure: Open flap debridement with a chemo-electric device + PRF — The defects will be removed from granulation tissue. Debridement by a chemical-electrical principle will be performed followed by application of PRF clots and membrane. Then, the flap will be closed and sutured.
  Arms: Open flap debridement with a chemo-electric device + PRF
Procedure: Open flap debridement with a chemo-electric device alone (control) — The defects will be removed from granulation tissue. Debridement by a chemical-electrical principle will be performed. Then the flap will be closed and sutured.
  Arms: Open flap debridement with a chemo-electric device alone

SUMMARY:
Platelet-rich fibrin (PRF) is a second-generation platelet concentrate used for tissue and bone regeneration. PRF releases growth factors such as TGF-β, PDGF, VEGF, IGF, and FGF, which are known to promote wound healing and bone regeneration. Thus, PRF may offer a promising therapeutic approach for peri-implantitis treatment. Numerous studies have reported beneficial effects of PRF on bone regeneration, bone augmentation, soft tissue healing, and ridge preservation. In infrabony periodontal defects, PRF has shown significant improvements in pocket depth reduction, clinical attachment level (CAL) gain, and bone fill.

However, a recent systematic review highlighted that evidence supporting PRF use in peri-implantitis remains limited, primarily due to a lack of adequately designed studies. Therefore, the aim of this project is to investigate whether PRF enhances regeneration in peri-implantitis defects. Specifically, it will assess whether surgical debridement of peri-implantitis defects-including electrochemical detoxification of implant surfaces using GalvoSurge-combined with PRF clot and membrane placement, improves treatment outcomes compared to surgical debridement and detoxification using GalvoSurge alone.

For this purpose, implants with peri-implantitis defects of comparable size will be randomly assigned to either the test or control group. After 12 months, implants will be clinically evaluated for radiographic defect fill, reduction in probing pocket depth (PPD), and bleeding on probing (BOP). The objective of this project is to verify, both radiographically and clinically, whether adjunctive PRF application enhances tissue regeneration and healing of peri-implantitis defects compared to open flap debridement (OFD) alone.

DETAILED DESCRIPTION:
Peri-implantitis is a chronic inflammatory condition around dental implants, associated with biofilm-mediated infection. The initial stage involves the formation of a bacterial biofilm in the peri-implant tissue, resulting in mucositis, which is characterized by erythema, bleeding, exudation, and swelling. With continued biofilm accumulation, mucositis can progress to peri-implantitis, which is marked by bone destruction. Due to varying definitions of peri-implantitis, the VIII European Workshop on Periodontology established diagnostic criteria, specifying progressive bone loss of ≥ 2 mm with clinical signs of inflammation. Recently, the American Academy of Periodontology and the European Federation of Periodontology suggested a threshold of ≥ 3 mm. Based on these definitions, recent meta-analyses have shown the prevalence of peri-implantitis to be approximately 18.5% at the patient level and 12.8% at the implant level, highlighting an increasingly significant problem within the global adult population.

Currently, treating peri-implantitis is challenging, costly, and often unpredictable. The primary goals of therapy are to resolve soft-tissue inflammation and stabilize the bony attachment. This requires effective removal of bacterial biofilms and deposits from implant surfaces to enable healing on a biologically clean surface. Peri-implantitis therapy often necessitates a surgical approach that includes surface decontamination with or without the use of a bone substitute. Despite these interventions, surgically treated cases demonstrate a high failure rate, with approximately 60% of cases showing recurrence, underscoring the need for innovative therapeutic approaches.

PRF has recently emerged as a viable alternative to recombinant growth factors due to its ability to support healing naturally. It is obtained by centrifuging blood to create a coagulated plasma that includes a complex mixture of growth factors within a fibrin network. This plasma can be further processed to extract a PRF membrane by squeezing out the serum. PRF membranes are increasingly used to enhance clinical outcomes by delivering growth factors at surgical sites, either alone or in combination with dental implants and collagen membranes.

This project aims to determine whether PRF enhances regeneration in peri-implantitis defects and to compare the outcomes of surgical debridement and implant detoxification combined with PRF clot and membrane placement, against debridement and detoxification alone. For this purpose, implants with peri-implantitis defects of comparable size will be randomly assigned to either the test or control group.

Study Endpoints:

Radiographic defect fill after one year, with a cut-off level of > 1.0 mm Clinical parameters: probing pocket depth (PPD), bleeding on probing (BoP), and keratinized tissue amount in mm on the oral and buccal implant sides Soft tissue healing as assessed by the Early Wound Healing Index by Wachtel Composite clinical index based on criteria established by Renvert et al. (2018) Patient-reported outcomes assessed through a visual analog scale

ELIGIBILITY:
Inclusion Criteria:

1. One or more peri-implant sites with PPD ≧ 5 mm combined with BOP/suppuration and
2. Peri-implant marginal bone loss, defined as a crater like defect ≧ 3 mm as assessed from intraoral radiographs
3. Good oral hygiene i.e. a plaque index <20%
4. Written informed consent

Exclusion Criteria:

1. History of chronic inflammatory disease
2. Severe systemic diseases
3. Medically confirmed diagnosis of diabetes mellitus
4. Anti-inflammatory prescription including prednisone
5. Smoking > 5 cigarettes
6. Pregnant or lactating women
7. < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — A balanced randomisation is being performed.
Enrollment: 40 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic defect fill after 12 months | Baseline, 12-month follow-up
  Radiographs of the implant will be made 12 months after the intervention and compared to baseline radiographs. Defect fill in mm will be assessed.

SECONDARY OUTCOMES:
Change of probing pocket depth | Baseline, 12-month follow-up
  Probing pocket depth (PPD) around the implants will be assessed at baseline and after 12 months after the intervention. PPD will be measured as the distance from the mucosal margin to the bottom of the peri-implant pocket using a periodontal probe with mm markings.
Change in bleeding on probing | Baseline, 12-month follow-up
  Bleeding on probing with 20 Ncm will be assessed at 6 sites around the implant at baseline and after 6 months. Bleeding on probing reflects the inflammatory state of the peri-implant tissues. Healthy peri-implant tissues present with no bleeding upon gentle probing. According to the grade of inflammation more sites around the implant bleed upon probing. 6 sites per implant will be assessed: mesiobuccal, midbuccal, distobuccal, distolingual, midlingual, mesiolingual. Change in the number of bleeding spots will be assessed from baseline to the 12-month follow-up.
Soft tissue healing | 2 days post-surgery, 7 days and 14 days post-surgery
  Healing during the first 2 weeks will be assessed by the early wound healing index. It is represented by a scale. When a low number on the scale is given, fast and uneventful healing occurs.
Radiographic and clinical composite index | Baseline, 12-month follow-up
  A composite outcome of no evidence of BoP (one site out of 6 will be accepted), with no suppuration at any site, PPD ≤ 5 mm and with ≥1 mm defect fill will be used for a successful outcome.
Patient-reported outcome pain assessed by visual analogue scale (VAS) | 2 days post-surgery, 7 days and 14 days post-surgery
  A 100 mm scale for pain will be used. Patient will be asked to mark their pain sensation with 0 representing no pain at all and 100 mm representing the worst imaginable pain. The time to recovery defined as pain <10 mm will be assessed.
Keratinized/attached tissue width | Baseline, 12-month follow-up
  The attached mucosa around an implant might be decisive for peri-implant health by facilitating oral hygiene. Keratinized tissue is mostly attached to the underlying bone. Keratinized tissue width will be measured as the distance from the mucosal margin to the border of the movable and lining mucosa. Lugol's solution will be used to discern the tissue border. The distance will be measured with a periodontal probe with mm markings. The keratinized/attached mucosa width will be measured at baseline and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Salvi, MD, Principal Investigator — University of Bern
Locations (1):
- Department of Periodontology, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Background] Bosshardt DD, Brodbeck UR, Rathe F, Stumpf T, Imber JC, Weigl P, Schlee M. Evidence of re-osseointegration after electrolytic cleaning and regenerative therapy of peri-implantitis in humans: a case report with four implants. Clin Oral Investig. 2022 Apr;26(4):3735-3746. doi: 10.1007/s00784-021-04345-1. Epub 2022 Mar 4. PMID 35244779
- [Background] Berglundh T, Lindhe J, Marinello C, Ericsson I, Liljenberg B. Soft tissue reaction to de novo plaque formation on implants and teeth. An experimental study in the dog. Clin Oral Implants Res. 1992 Mar;3(1):1-8. doi: 10.1034/j.1600-0501.1992.030101.x. PMID 1420721
- [Background] Derks J, Tomasi C. Peri-implant health and disease. A systematic review of current epidemiology. J Clin Periodontol. 2015 Apr;42 Suppl 16:S158-71. doi: 10.1111/jcpe.12334. PMID 25495683
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part III: leucocyte activation: a new feature for platelet concentrates? Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e51-5. doi: 10.1016/j.tripleo.2005.07.010. PMID 16504851
- [Background] Roccuzzo M, Layton DM, Roccuzzo A, Heitz-Mayfield LJ. Clinical outcomes of peri-implantitis treatment and supportive care: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:331-350. doi: 10.1111/clr.13287. PMID 30328195
- [Background] Lang NP, Bragger U, Walther D, Beamer B, Kornman KS. Ligature-induced peri-implant infection in cynomolgus monkeys. I. Clinical and radiographic findings. Clin Oral Implants Res. 1993 Mar;4(1):2-11. doi: 10.1034/j.1600-0501.1993.040101.x. PMID 8329533
- [Background] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729
- [Background] Pontoriero R, Tonelli MP, Carnevale G, Mombelli A, Nyman SR, Lang NP. Experimentally induced peri-implant mucositis. A clinical study in humans. Clin Oral Implants Res. 1994 Dec;5(4):254-9. doi: 10.1034/j.1600-0501.1994.050409.x. PMID 7640340
- [Background] Pradeep AR, Karvekar S, Nagpal K, Patnaik K, Raju A, Singh P. Rosuvastatin 1.2 mg In Situ Gel Combined With 1:1 Mixture of Autologous Platelet-Rich Fibrin and Porous Hydroxyapatite Bone Graft in Surgical Treatment of Mandibular Class II Furcation Defects: A Randomized Clinical Control Trial. J Periodontol. 2016 Jan;87(1):5-13. doi: 10.1902/jop.2015.150131. Epub 2015 Oct 5. PMID 26439386
- [Result] Hamzacebi B, Oduncuoglu B, Alaaddinoglu EE. Treatment of Peri-implant Bone Defects with Platelet-Rich Fibrin. Int J Periodontics Restorative Dent. 2015 May-Jun;35(3):415-22. doi: 10.11607/prd.1861. PMID 25909530